CLINICAL TRIAL: NCT04200417
Title: Phase I Study of Transarterial Chemoembolization of Lung Metastases
Brief Title: Chemoembolization for Lung Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-371
Record Dates: First submitted 2019-12-13; First posted 2019-12-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2022-04

CONDITIONS: Lung Metastases; Endobronchial Metastases; Pleural Metastases; Mediastinal Metastases
Keywords: Unresectable Lung Cancer; Unresectable Endobronchial Mestastases; Unresectable Pleural Metastases; Unresectable Mediastinal Metastases; Lung Chemoembolization; 19-371; Memorial Sloan Kettering Cancer Center
MeSH Terms: interventions — Chemoembolization, Therapeutic; Mitomycin; Ethiodized Oil; trisacryl gelatin microspheres

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lung, Endobronchial, Mediastinal or Pleural Metastases (Experimental): Participants will have unresectable and unablatable lung, endobronchial, mediastinal, or pleural metastases (from any primary) that are not responding to chemotherapy
  Interventions: Procedure: Chemoembolization; Drug: Mitomycin C; Drug: Lipiodol; Drug: Embospheres

INTERVENTIONS:
Procedure: Chemoembolization — Chemoembolization will be performed via the artery (bronchial, non-bronchial systemic, or pulmonary) that shows the greatest tumor enhancement on angiography. Chemoembolization will be performed using a lipiodol / mitomycin emulsion, followed by spherical particles.
Drug: Mitomycin C — Mitomycin (5mg/m^2,maximum mitomycin dose 20 mg) will be dissolved in lipiodol at 2 mg/ml on the day of procedure.
Drug: Lipiodol — Mitomycin (5mg/m^2,maximum mitomycin dose 20 mg) will be dissolved in lipiodol at 2 mg/ml on the day of procedure.
Drug: Embospheres — Embospheres are non-resorbable spherical microspheres (trisacryl gelatin) that are FDA-approved for embolization of hypervascular tumors.

SUMMARY:
This study is being done to determine if it is safe to perform lung chemoembolization and if the lung chemoembolization procedure can successfully deliver chemotherapy to lung tumors.

ELIGIBILITY:
Inclusion Criteria:

* Lung, endobronchial, pleural, or mediastinal metastases that are not responding to systemic chemotherapy, and that are not amenable to ablation, resection, or SBRT.
* At least 18 years old.
* ECOG performance status 0 or 1

Exclusion Criteria:

* Primary lung cancer
* >50% of a lung is replaced with tumor
* Oxygen saturation <92% on room air
* FEV1 <60%
* Pulmonary hypertension (diagnosed or suspected on echocardiography, CT, MRI, or direct pressure measurement)
* Recent pulmonary embolism (within 3 months)
* Pulmonary arteriovenous malformation
* Active lung infection (pneumonia, empyema, or lung abscess requiring therapy within 1 month)
* Symptomatic heart failure (dyspnea, volume overload)
* Left bundle branch block (contraindication to pulmonary angiography)
* Renal failure (eGFR <30 mL/min/1.73m^2)
* Pregnancy
* Breastfeeding
* Altered mental status that would interfere with consent or follow-up
* Platelets < 100,000 (after transfusion, if needed)
* INR>2 (after transfusion, if needed)
* Hemoglobin <7 (after transfusion, if needed)
* Hyperthyroidism (contraindication to lipiodol)
* Planned radioactive iodine imaging or therapy (contraindication to lipiodol)
* Allergy to lipiodol or mitomycin
* Allergy to iodinated contrast that can not be treated with steroid / diphenhydramine premedication
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Participant toxicity will be evaluated according to CTCAE v5.0 | Up to 12 months post treatment
  Safety will be evaluated by participant toxicity according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Solomon, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memoral Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack (Consent Only), Commack, New York
  - Memoral Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org